CLINICAL TRIAL: NCT01282502
Title: Phase I Study of Chemoradiation With Midostaurin (PKC412) For Locally Advanced Rectal Cancer
Brief Title: Midostaurin (PKC412) for Locally Advanced Rectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Theodore Sunki Hong, Radiation Oncologist, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-457
Record Dates: First submitted 2011-01-21; First posted 2011-01-25 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Adenocarcinoma of the Rectum
Keywords: rectal cancer; chemotherapy; chemoradiation
MeSH Terms: conditions — Rectal Neoplasms | interventions — midostaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Midostaurin with chemoradiation (Experimental)
  Interventions: Drug: Midostaurin

INTERVENTIONS:
Drug: Midostaurin — 50 mg BID for 8 cycles

SUMMARY:
This study combines midostaurin (PKC412) with radiation and a standard chemotherapy drug call 5-Fluorouracil (5-FU) for subjects with advanced rectal cancer. Midostaurin is a type of kinase inhibitor which works by blocking proteins associated with cancer cell growth. Previous studies also suggest that midostaurin may help increase the effectiveness of radiation therapy. In this research we are looking for the highest dose of midostaurin that can be given safely in combination with standard chemoradiation.

DETAILED DESCRIPTION:
Midostaurin capsules will be taken by mouth for 8 weeks. For the first 2 weeks midostaurin will be taken alone (no chemoradiation). After 2 weeks standard chemoradiation will be added to the midostaurin regimen. Subjects receive midostaurin and chemoradiation for an additional 6 weeks. Physical exams will be done weekly. Blood samples will be taken and an optional tumor biopsy will be performed in week 2.

4-5 weeks after completing chemoradiation and midostaurin subjects will undergo surgery as standard of care. Tumor tissue from the surgery will be used for research purposes. A Ct scan of chest, abdomen, and pelvis will be performed.

After completion of surgery, subjects will have an end of study visit with physical exam, blood tests. CT scans of chest, abdomen, and pelvis will be performed yearly for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the rectum
* T3/4 or N+ disease
* Life expectancy > 3 months
* Normal organ and marrow function

Exclusion Criteria:

* Metastatic disease
* Pregnant or breastfeeding
* Prior radiotherapy
* Receiving other investigational agents
* History of inflammatory bowel disease
* Active scleroderma or CREST syndrome
* Uncontrolled intercurrent illness
* History of a different malignancy unless disease free for at least 5 years
* HIV or active viral hepatitis
* Impaired cardiac function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-08; Primary Completion 2015-03 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
To determine Maximum Tolerated Dose (MTD) of midostaurin in combination with standard 5-FU chemoradiation | 1.5 years

SECONDARY OUTCOMES:
To determine the rate of Dworak Tumor Regression Grade 3/4 for locally advanced rectal cancer treated with study combination at the MTD, stratified by KRAS status (mutant vs. wild type) | 1.5 years
To determine surgical complication rate in patients who received preoperative radiation therapy | 1.5 years
Perform an exploratory analysis of the impact of selected mutations in APC, PTEN, BRAF, NRAS, and PIK3CA, among other genes | 1.5 year
To evaluate proteomic markers of response and resistance to midostaurin-based chemoradiation | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Theodore S Hong, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts